CLINICAL TRIAL: NCT05938257
Title: Comparative Study Between Arthroscopic Versus Open Surgical Discopexy for Treatment of Temporomandibular Joint Anterior Disc Displacement Without Reduction (RCT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Gamal Thabet (Other)
Responsible Party: Sponsor-Investigator, Mohamed Gamal Thabet, Assiut university, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mohamed G Thabet
Record Dates: First submitted 2023-06-20; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Efficacy of TMJ Arthroscopy

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TMJ dysfunction (Experimental): TMJ discopexy
  Interventions: Procedure: TMJ discopexy

INTERVENTIONS:
Procedure: TMJ discopexy — Arthroscopic versus open TMJ discopexy

SUMMARY:
Temporomandibular joint dysfunction (TMD) represents a common health problem. A recent systematic review and meta-analysis in 2021 concluded that the prevalence of TMD was 31% for adults and 11% for adolescence.

Many believe that TMD symptoms are related to internal derangement of the temporomandibular joint (TMJ), which is usually in the form of anterior disc displacement(ADD) and it is often associated with pain, clicking, limited range of motion, and even osteoarthritic changes.

Treatment of TMD include non-surgical and surgical modalities. Non-surgical treatment includes instructions, pharmacotherapy, occlusal splints and physiotherapy. Patients who do not respond to non-surgical therapy may require surgical interventions that include minimally invasive procedures (arthroscopy and arthrocentesis) and open surgery.

Arthroscopy of the TMJ was first introduced by Ohnishi in 1975, it involves lysis of adhesions and lavage of the superior joint space, as well as repositioning of a displaced disc.

Open TMJ surgery can be very effective at eliminating symptoms of pain, limited mouth opening and mandibular dysfunction.

DETAILED DESCRIPTION:
Patients are assigned randomly into two groups; group (1) for arthroscopic discopexy, and group (2) for open discopexy.

History taking: personal history; name, age, gender and occupation. Patient's complaint(s); as TMJ clicking, pain, locking and limited mouth opening.

Clinical examination: for TMJ clicking and tenderness, measurement of maximum inter-incisal opening (MIO) in mm. Examination of facial symmetry, dental occlusion and dentoskeletal deformity.

Radiological evaluation: Computed Tomography (CT) scan of maxillofacial bones. Magnetic Resonance Imaging (MRI) for TMJ, to confirm anterior disc displacement without reduction.

Operative procedures: will be carried out by the same team, under general anaesthesia, nasotracheal intubation and supine position.

Group (1) for arthroscopic discopexy: using 1.9 mm diameter - 30-degree scope. The procedure is performed through three ports and a suture-passing spinal needle 18 gauge. One port for the scope, second port for manipulation and reduction of the displaced disc and third port for retrieval of the suture used for discopexy. The suture used is 2-0 polypropylene, which is tied down in the extra-capsular tissue.

Group (2) for open discopexy: through pre-auricular incision. Exposure of the temporomandibular joint capsule, incision is made through the lateral capsule into the superior joint space and the disc is repositioned. Discopexy is done using 2-0 polypropylene suture.

Follow up will be at intervals of 1, 3, 6 and 12 months after the operation for clinical assessment of pain by Visual Analogue Scale (VAS), MIO in mm, joint clicking and complications.

MRI of TMJ is performed after one month of surgery to evaluate position of the articular disc.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TMD in the form of anterior disc displacement without reduction
* Age: 20 - 50 years' old

Exclusion Criteria:

* Secondary TMD
* TMJ ankylosis
* Structural deformity of TMJ
* Previous surgical intervention to TMJ
* Patients who are unfit for surgery

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
TMJ pain | one year
  change of pain on a visual analogue scale from 0 to 10 with decreased number means less pain

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Government, Egypt